CLINICAL TRIAL: NCT02393859
Title: Phase 3 Trial to Investigate the Efficacy, Safety, and Tolerability of Blinatumomab as Consolidation Therapy Versus Conventional Consolidation Chemotherapy in Pediatric Subjects With HR First Relapse B-precursor ALL
Brief Title: Phase 3 Trial of Blinatumomab vs Standard Chemotherapy in Pediatric Subjects With HIgh-Risk (HR) First Relapse B-precursor Acute Lymphoblastic Leukemia (ALL)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20120215; 2014-002476-92 (EudraCT Number)
Record Dates: First submitted 2015-03-16; First posted 2015-03-20 (Estimated); Results first posted 2020-07-13 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Leukemia, Acute Lymphoblastic
Keywords: ALL; High-risk first relapse B-precursor ALL; Precursor Cell Lymphoblastic Leukemia; Neoplasms; Lymphoproliferative Disorders; Immunoproliferative Disorders; Antibodies, Bispecific
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasms; Lymphoproliferative Disorders; Immunoproliferative Disorders | interventions — blinatumomab; Dexamethasone; Daunorubicin; Methotrexate; Ifosfamide; pegaspargase; asparaginase erwinia chrysanthemi recombinant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High Risk Consolidation 3 (HC3) Chemotherapy (Active Comparator): One week of treatment with HC3 followed by 3 weeks of no treatment. The standard intensive consolidation chemotherapy course HC3 includes dexamethasone (10 mg/m^2/day intravenous [IV] on Days 1-6), vincrisitne (1.5 mg/m^2/day IV on Days 1 and 6), daunorubicin (30 mg/m^2 IV over 24 hours on Day 5), methotrexate (1 g/m^2 IV over 36 hours on Day 1), ifosfamide (800 mg/m^2 IV for 1 hour on Days 2-4), and pegylated [PEG]-asparaginase (1000 U/m^2 IV for 2 hours or intramuscularly [IM] on Day 6) or, if allergic, erwinia-asparaginase (20,000 units/m^2 IV or IM every 48 hours for a total of 6 doses).
  Interventions: Drug: Dexamethasone; Drug: Vincrisitne; Drug: Daunorubicin; Drug: Methotrexate; Drug: Ifosfamide; Drug: PEG-asparaginase; Drug: Erwinia-asparaginase
- Blinatumomab (Experimental): 15 μg/m^2/day as a continuous intravenous infusion (CIVI) for 4 weeks
  Interventions: Drug: Blinatumomab

INTERVENTIONS:
Drug: Blinatumomab — 15 μg/m^2/day as a continuous intravenous infusion (CIVI) for 4 weeks
  Other Names: Blincyto, AMG103
  Arms: Blinatumomab
Drug: Dexamethasone — 10 mg/m^2/day intravenous (IV) on Days 1-6
  Arms: High Risk Consolidation 3 (HC3) Chemotherapy
Drug: Vincrisitne — 1.5 mg/m^2/day IV on Days 1 and 6
  Arms: High Risk Consolidation 3 (HC3) Chemotherapy
Drug: Daunorubicin — 30 mg/m^2 IV over 24 hours on Day 5
  Arms: High Risk Consolidation 3 (HC3) Chemotherapy
Drug: Methotrexate — 1 g/m^2 IV over 36 hours on Day 1
  Arms: High Risk Consolidation 3 (HC3) Chemotherapy
Drug: Ifosfamide — 800 mg/m^2 IV for 1 hour on Days 2-4
  Arms: High Risk Consolidation 3 (HC3) Chemotherapy
Drug: PEG-asparaginase — 1000 U/m^2 IV for 2 hours or intramuscularly (IM) on Day 6
  Arms: High Risk Consolidation 3 (HC3) Chemotherapy
Drug: Erwinia-asparaginase — In case of allergic reaction to PEG-asparaginase, participants could change to erwinia-asparaginase, 20,000 units/m2 every 48 hours for a total of 6 doses
  Arms: High Risk Consolidation 3 (HC3) Chemotherapy

SUMMARY:
B-precursor ALL is an aggressive malignant disease. Therapy is usually stratified according to risk characteristics to ensure that appropriate treatment is administered to patients with high-risk of relapse. In general, pediatric treatment regimens are more intense than those employed in adults and include courses of combination chemotherapy. Standard of care chemotherapy is associated with considerable toxicity. There is a lack of novel treatment options for subjects who relapse or are refractory to treatment. Therefore, innovative therapeutic approaches are urgently needed. Blinatumomab is a bispecific single-chain antibody construct designed to link B cells and T cells resulting in T cell activation and a cytotoxic T cell response against CD19 expressing cells. This study will evaluate the event-free survival (EFS) after treatment with blinatumomab when compared to standard of care (SOC) chemotherapy. The effect of blinatumomab on overall survival and reduction of minimal residual disease compared to SOC chemotherapy will also be investigated.

DETAILED DESCRIPTION:
Patients will be randomized in a 1:1 ratio to receive either one cycle of blinatumomab or one block of standard high-risk consolidation chemotherapy. Blinatumomab is administered as a continuous intravenous infusion (CIVI). One cycle of blinatumomab treatment includes 4 weeks of CIVI of blinatumomab. After completing consolidation therapy, the patients should undergo alloHSCT depending on their bone marrow status. The patients will be followed up until the last subject on study is 36 months following alloHSCT or has died, whichever is first.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Philadelphia chromosome negative (Ph-) high-risk (HR) first relapse B-precursor acute lymphoblastic leukemia (ALL; as defined by International Berlin-Frankfurt-Muenster study group/International study for treatment of childhood relapsed ALL [I-BFM SG/IntReALL] criteria)
* Subjects with bone marrow blast percentage < 5% (M1) or bone marrow blast percentage < 25% and ≥5% (M2) marrow at the time of randomization,
* Age > 28 days and < 18 years at the time of informed consent/assent
* Subject's legally acceptable representative has provided informed consent when the subject is legally too young to provide informed consent and the subject has provided written assent based on local regulations and/or guidelines prior to any study-specific activities/procedures being initiated
* Availability of the following material from relapse diagnosis for central analysis of minimal residual disease (MRD) by polymerase chain reaction (PCR): clone-specific primers and reference deoxyribonucleic acid (DNA), as well as primer sequences and analyzed sequences of clonal rearrangements (cases with isolated extramedullary relapse or cases with technical and/or logistic hurdles to obtain and process bone marrow material are exempt from providing this material. In these cases, central MRD analysis only by Flow is permitted).

Exclusion Criteria:

* Clinically relevant central nervous system (CNS) pathology requiring treatment (eg, unstable epilepsy). Evidence of current CNS (CNS 2, CNS 3) involvement by ALL. Subjects with CNS relapse at the time of relapse are eligible if CNS is successfully treated prior to enrollment
* Peripheral neutrophils < 500/μL prior to start of treatment
* Peripheral platelets < 50,000/μL prior to start of treatment
* Currently receiving treatment in another investigational device or drug study or less than 4 weeks since ending treatment on another investigational device or drug study(s), procedures required by IntReALL high-risk (HR) guidelines are allowed
* Chemotherapy related toxicities that have not resolved to ≤ grade 2 (except for parameters defined in Exclusion Criteria 202, 203, 204, and 217)
* Symptoms and/or clinical signs and/or radiological and/or sonographic signs that indicate an acute or uncontrolled chronic infection, any other concurrent disease or medical condition that could be exacerbated by the treatment or would seriously complicate compliance with the protocol
* Abnormal renal or hepatic function prior to start of treatment (day 1) as defined below
* Abnormal serum creatinine based on age/gender
* Total bilirubin > 3.0 mg/dL prior to start of treatment (unless related to Gilbert's or Meulengracht disease)
* Documented infection with human immunodeficiency virus (HIV)
* Known hypersensitivity to immunoglobulins or any of the products or components to be administered during dosing (excluding asparaginase)
* Post-menarchal female subject who is pregnant or breastfeeding, or is planning to become pregnant or breastfeed while receiving protocol-specified therapy and for at least 12 months after the last dose of chemotherapy
* Post-menarchal female subject who is not willing to practice true sexual abstinence or use a highly effective form of contraception while receiving protocol-specified therapy and for at least 12 months after the last dose of chemotherapy
* Sexually mature male subject who is not willing to practice true sexual abstinence or use a condom with spermicide while receiving protocol-specified therapy and for at least 6 months after last dose of chemotherapy. In countries where spermicide is not available, a condom without spermicide is acceptable
* Sexually mature male subject who is not willing to abstain from sperm donation while receiving protocol-specified therapy and for at least 6 months after last dose of chemotherapy
* Subject likely to not be available to complete all protocol-required study visits or procedures, including follow-up visits, and/or to comply with all required study procedures to the best of the subject's and investigator's knowledge
* History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion
* Placed into an institution due to juridical or regulatory ruling.

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 111 (Actual)
Dates: Start 2015-11-10 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2022-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (97):
- Research Site, Ciudad Autonoma de Buenos Aires, Buenos Aires, Argentina
- Australia (4):
  - Research Site, Randwick, New South Wales
  - Research Site, Westmead, New South Wales
  - Research Site, South Brisbane, Queensland
  - Research Site, Parkville, Victoria
- Austria (3):
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Vienna
- Belgium (4):
  - Research Site, Brussels
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Liège
- Brazil (3):
  - Research Site, Curitba, Paraná
  - Research Site, Porto Alegre, Rio Grande do Sul
  - Research Site, São Paulo, São Paulo
- Research Site, Prague, Czechia
- Research Site, København Ø, Denmark
- France (9):
  - Research Site, Bordeaux
  - Research Site, Lille
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Strasbourg
  - Research Site, Vandœuvre-lès-Nancy
- Germany (16):
  - Research Site, Berlin
  - Research Site, Düsseldorf
  - Research Site, Erlangen
  - Research Site, Essen
  - Research Site, Frankfurt am Main
  - Research Site, Freiburg im Breisgau
  - Research Site, Giessen
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Jena
  - Research Site, Kiel
  - Research Site, München
  - Research Site, Münster
  - Research Site, Tübingen
  - Research Site, Ulm
  - Research Site, Würzburg
- Research Site, Goudi, Greece
- Israel (5):
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Petah Tikva
  - Research Site, Tel Aviv
  - Research Site, Tel Litwinsky
- Italy (8):
  - Research Site, Bologna
  - Research Site, Genova
  - Research Site, Monza (MB)
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Pavia
  - Research Site, Roma
  - Research Site, Torino
- Mexico (3):
  - Research Site, Guadalajara, Jalisco
  - Research Site, Mexico City, Mexico City
  - Research Site, Monterrey, Nuevo León
- Netherlands (2):
  - Research Site, Rotterdam
  - Research Site, Utrecht
- Research Site, Oslo, Norway
- Poland (5):
  - Research Site, Bydgoszcz
  - Research Site, Krakow
  - Research Site, Lublin
  - Research Site, Wroclaw
  - Research Site, Zabrze
- Portugal (2):
  - Research Site, Lisbon
  - Research Site, Porto
- Romania (2):
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
- Russia (2):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- Spain (9):
  - Research Site, Málaga, Andalusia
  - Research Site, Seville, Andalusia
  - Research Site, Santander, Cantabria
  - Research Site, Barcelona, Catalonia
  - Research Site, Santiago de Compostela, Galicia
  - Research Site, Boadilla del Monte, Madrid
  - Research Site, El Palmar, Murcia
  - Research Site, Valencia, Valencia
  - Research Site, Madrid
- Research Site, Stockholm, Sweden
- Switzerland (2):
  - Research Site, Basel
  - Research Site, Zurich
- Turkey (Türkiye) (4):
  - Research Site, Adana
  - Research Site, Antalya
  - Research Site, Izmir
  - Research Site, Kayseri
- United Kingdom (8):
  - Research Site, Birmingham
  - Research Site, Bristol
  - Research Site, Glasgow
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Newcastle upon Tyne
  - Research Site, Sheffield
  - Research Site, Sutton

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Locatelli F, Eckert C, Hrusak O, Buldini B, Sartor M, Zugmaier G, Zeng Y, Pilankar D, Morris J, von Stackelberg A. Blinatumomab overcomes poor prognostic impact of measurable residual disease in pediatric high-risk first relapse B-cell precursor acute lymphoblastic leukemia. Pediatr Blood Cancer. 2022 Aug;69(8):e29715. doi: 10.1002/pbc.29715. Epub 2022 Apr 28. PMID 35482538
- [Background] Blinatumomabe em pacientes pediátricos com leucemia linfoblástica aguda B em primeira recidiva de alto risco: um estudo de custo-efetividade. van Beurden-Tan CHY, Ribeiro RA, Seber A, de Martino Lee ML, Marçola M, Schuetz R, Loggetto SR, Maiolino A. Jornal Brasileiro de Economia da Saúde 14(1): 41-50. 10.21115/JBES.v14.n1.p41-50
- [Background] Locatelli F, Zugmaier G, Rizzari C, Morris JD, Gruhn B, Klingebiel T, Parasole R, Linderkamp C, Flotho C, Petit A, Micalizzi C, Mergen N, Mohammad A, Kormany WN, Eckert C, Moricke A, Sartor M, Hrusak O, Peters C, Saha V, Vinti L, von Stackelberg A. Effect of Blinatumomab vs Chemotherapy on Event-Free Survival Among Children With High-risk First-Relapse B-Cell Acute Lymphoblastic Leukemia: A Randomized Clinical Trial. JAMA. 2021 Mar 2;325(9):843-854. doi: 10.1001/jama.2021.0987. PMID 33651091
- [Background] Caillon M, Brethon B, van Beurden-Tan C, Supiot R, Le Mezo A, Chauny JV, Majer I, Petit A. Cost-Effectiveness of Blinatumomab in Pediatric Patients with High-Risk First-Relapse B-Cell Precursor Acute Lymphoblastic Leukemia in France. Pharmacoecon Open. 2023 Jul;7(4):639-653. doi: 10.1007/s41669-023-00411-4. Epub 2023 Apr 18. PMID 37071263
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 48 centers across 13 countries (Europe, Australia, Israel). The first participant was enrolled on 10 November 2015. The last participant enrolled on 30 August 2019.
  The primary completion date was 17 July 2019 and the study completion date was 21 November 2022.
Pre-assignment Details: After a 3-week screening period, participants were enrolled and randomized 1:1 into 1 of 2 treatment groups: High Risk Consolidation 3 (HC3) chemotherapy or blinatumomab.
  Randomization was stratified by age and bone marrow/minimal residual disease (MRD) status.
Groups:
- HC3 Chemotherapy: One week of treatment with HC3 followed by 3 weeks of no treatment. The standard intensive consolidation chemotherapy course HC3 includes dexamethasone (10 mg/m^2/day intravenous [IV] on Days 1-6), vincrisitne (1.5 mg/m^2/day IV on Days 1 and 6), daunorubicin (30 mg/m^2 IV over 24 hours on Day 5), methotrexate (1 g/m^2 IV over 36 hours on Day 1), ifosfamide (800 mg/m^2 IV for 1 hour on Days 2-4), and pegylated [PEG]-asparaginase (1000 U/m^2 IV for 2 hours or intramuscularly [IM] on Day 6) or, if allergic, erwinia-asparaginase (20,000 units/m^2 IV or IM every 48 hours for a total of 6 doses).
- Blinatumomab: One 4-week cycle of blinatumomab 15 μg/m^2/day as a continuous intravenous infusion (CIVI).
Period: Overall Study
Arm/Group | HC3 Chemotherapy | Blinatumomab
Started | 57 | 54
Participants Treated | 52 | 54
Participants in the Primary Analysis Population (Included all randomized participants analyzed according to their randomized treatment assignment, regardless of treatment received (the full analysis set; FAS) at the primary completion date (17 July 2019)) | 54 | 54
Participants in the Final Analysis Population (Included all randomized participants analyzed according to their randomized treatment assignment, regardless of treatment received (FAS) at study completion (21 November 2022)) | 57 | 54
Completed | 16 | 33
Not Completed | 41 | 21
Not completed — Decision by Sponsor | 2 | 4
Not completed — Withdrawal by Subject | 11 | 6
Not completed — Death | 27 | 10
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: The FAS included all randomized participants analyzed according to their randomized treatment assignment, regardless of the treatment received.
Groups:
- HC3 Chemotherapy: One week of treatment with HC3 followed by 3 weeks of no treatment. The standard intensive consolidation chemotherapy course HC3 includes dexamethasone (10 mg/m^2/day IV on Days 1-6), vincrisitne (1.5 mg/m^2/day IV on Days 1 and 6), daunorubicin (30 mg/m^2 IV over 24 hours on Day 5), methotrexate (1 g/m^2 IV over 36 hours on Day 1), ifosfamide (800 mg/m^2 IV for 1 hour on Days 2-4), and pegylated [PEG]-asparaginase (1000 U/m^2 IV for 2 hours or IM on Day 6) or, if allergic, erwinia-asparaginase (20,000 units/m^2 IV or IM every 48 hours for a total of 6 doses).
- Total: Total of all reporting groups
Arm/Group | HC3 Chemotherapy | Blinatumomab | Total
Number analyzed (Participants) | 57 | 54 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.6 (4.3) | 7.3 (4.4) | 7.0 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 24 | 58
  Male | 23 | 30 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 54 | 53 | 107
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 46 | 50 | 96
  Other, Not Specified | 5 | 3 | 8
  Asian | 3 | 1 | 4
  Black or African American | 3 | 0 | 3
Stratification Factor: Age Category [Count of Participants; unit: Participants]
  1 to 9 years | 41 | 39 | 80
  Other (< 1 year and > 9 years) | 16 | 15 | 31
Stratification Factor: Marrow/Minimal Residual Disease (MRD) [Number; unit: participants] — M1: representative bone marrow aspirate or biopsy with blasts < 5%, with satisfactory cellularity and with regenerating hematopoiesis; M2: representative bone marrow aspirate or biopsy with ≥ 5% and < 25% blasts; MRD=minimal residual disease levels ≥ 10^-3 or < 10^-3, by polymerase chain reaction (PCR) or flow cytometry.
  participants
    M1 Marrow + MRD level ≥ 10^-3 | 17 | 15 | 32
    M1 Marrow + MRD level < 10^-3 | 36 | 35 | 71
    M2 Marrow | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Kaplan Meier Estimate: Event-Free Survival (EFS; Primary Analysis)
Description: EFS is calculated from the time of randomization until the date of relapse or M2 marrow (representative bone marrow aspirate or biopsy with ≥ 5% and < 25% blasts) after having achieved a complete remission (CR), failure to achieve a CR at the end of treatment, second malignancy, or death due to any cause, whichever occurs first. Participants who failed to achieve a CR following treatment with investigational product (IP) or who died before the disease assessment at the end of treatment were considered treatment failures and assigned an EFS duration of 1 day. Participants still alive and event-free were censored on their last disease assessment date.
  Participants were said to be in CR when they had the following:
  * M1 marrow
  * Peripheral blood without blasts
  * Absence of extramedullary leukemic involvement
  Months are calculated as days from randomization date to event/censor date, divided by 30.5.
Time Frame: As of the primary analysis data cutoff date (17 July 2019), overall median follow-up time for EFS was 22.4 months.
Population: Full Analysis Set: randomized participants analyzed according to their randomized treatment assignment, regardless of the treatment received (primary analysis population).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | HC3 Chemotherapy | Blinatumomab
Number analyzed (Participants) | 54 | 54
months | 7.4 [4.5 to 12.7] | NA [12.0 to NA] — NA=not estimable (median EFS and upper confidence interval [CI] were not reached at time of data cutoff)
Statistical Analysis 1: Comparison: HC3 Chemotherapy vs Blinatumomab; Test type: Superiority; p < 0.001, Stratified log-rank test — Stratification factors were: age (1 to 9 years vs other [< 1 year and > 9 years]), and marrow/MRD status (M1 with MRD level < 10^-3 vs M1 with MRD level ≥ 10^-3 vs M2); Normal score = -11.54 — A normal score < 0 indicates fewer than expected events for blinatumomab relative to HC3 and therefore a longer event-free survival time
Statistical Analysis 2: Comparison: HC3 Chemotherapy vs Blinatumomab; Test type: Superiority; p = 0.001, Unstratified log-rank test; Normal score = -11.16 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: HC3 Chemotherapy vs Blinatumomab; Test type: Superiority; Stratified hazard ratio (HR) = 0.36, 95% CI 2-sided [0.19 to 0.66] — Cox proportional hazard model. Stratification factors were: age and marrow/MRD status. (HR < 1.0 indicates a lower average event rate and a longer EFS for blinatumomab relative to HC3.)
Statistical Analysis 4: Comparison: HC3 Chemotherapy vs Blinatumomab; Test type: Superiority; Unstratified HR = 0.39, 95% CI 2-sided [0.22 to 0.70] — Cox proportional hazard model. (HR < 1.0 indicates a lower average event rate and a longer EFS for blinatumomab relative to HC3.)
Statistical Analysis 5: Comparison: HC3 Chemotherapy vs Blinatumomab; Test type: Superiority; Stratified HR w/time-dependent covariate = 0.36, 95% CI 2-sided [0.20 to 0.64] — Cox proportional hazard model including time from randomization to allogeneic hematopoietic stem cell transplant. Stratification factors: age and marrow/MRD status. (HR <1.0=lower average event rate and longer EFS for blinatumomab relative to HC3.)

2. Primary Outcome: Kaplan Meier Estimate: EFS (Final Analysis)
Description: EFS is calculated from the time of randomization until the date of relapse or M2 marrow after having achieved a CR, failure to achieve a CR at the end of treatment, second malignancy, or death due to any cause, whichever occurs first. Participants who failed to achieve a CR following treatment with IP or who died before the disease assessment at the end of treatment were considered treatment failures and assigned an EFS duration of 1 day. Participants still alive and event-free were censored on their last disease assessment date.
  Participants were said to be in CR when they had the following:
  * M1 marrow
  * Peripheral blood without blasts
  * Absence of extramedullary leukemic involvement
  Months are calculated as days from randomization date to event/censor date, divided by 30.5.
Time Frame: At final analysis, overall median follow-up time for EFS was 51.9 months.
Population: FAS: randomized participants analyzed according to their randomized treatment assignment, regardless of the treatment received (final analysis population).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | HC3 Chemotherapy | Blinatumomab
Number analyzed (Participants) | 57 | 54
months | 7.8 [5.8 to 13.4] | NA [24.8 to NA] — Median and upper 95% CI were not estimable due to too few events.
Statistical Analysis 1: Comparison: HC3 Chemotherapy vs Blinatumomab; Test type: Superiority; p < 0.001, Stratified log-rank test — [p-value comment as in outcome 1, analysis 1]; Normal score = -13.90 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: HC3 Chemotherapy vs Blinatumomab; Test type: Superiority; p < 0.001, Unstratified log-rank test; Normal score = -13.61 — A normal score < 0 indicates fewer than expected events for Blinatumomab relative to HC3 and therefore a longer event free survival time
Statistical Analysis 3: Comparison: HC3 Chemotherapy vs Blinatumomab; Test type: Superiority; Stratified HR = 0.35, 95% CI 2-sided [0.20 to 0.61] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: HC3 Chemotherapy vs Blinatumomab; Test type: Superiority; Unstratified HR = 0.38, 95% CI 2-sided [0.22 to 0.65] — [estimate comment as in outcome 1, analysis 4]
Statistical Analysis 5: Comparison: HC3 Chemotherapy vs Blinatumomab; Test type: Superiority; Stratified HR w/time-dependent covariate = 0.34, 95% CI 2-sided [0.20 to 0.59] — [estimate comment as in outcome 1, analysis 5]

3. Secondary Outcome: Kaplan Meier Estimate: Overall Survival (OS)
Description: OS was calculated from time of randomization until death due to any cause. Participants still alive were censored at the date they were last known to be alive.
  Months were calculated as days from randomization date to event/censor date, divided by 30.5.
Time Frame: At final analysis, overall median follow-up time for OS was 55.2 months.
Population: FAS: randomized participants analyzed according to their randomized treatment assignment, regardless of the treatment received.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | HC3 Chemotherapy | Blinatumomab
Number analyzed (Participants) | 57 | 54
months | 25.6 [17.5 to NA] — Upper 95% CI was not estimable due to too few events. | NA [NA to NA] — Median and 95% CIs were not estimable due to too few events.
Statistical Analysis 1: Comparison: HC3 Chemotherapy vs Blinatumomab; Test type: Superiority; p = 0.001, Stratified log-rank test — [p-value comment as in outcome 1, analysis 1]; Normal score = -10.14 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: HC3 Chemotherapy vs Blinatumomab; Test type: Superiority; p < 0.001, Unstratified log-rank test; Normal score = -10.32 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: HC3 Chemotherapy vs Blinatumomab; Test type: Superiority; Stratified HR = 0.33, 95% CI 2-sided [0.16 to 0.66] — Cox proportional hazard model. Stratification factors were: age and marrow/MRD status. (HR < 1.0 indicates a lower average event rate and a longer survival for blinatumomab relative to HC3.)
Statistical Analysis 4: Comparison: HC3 Chemotherapy vs Blinatumomab; Test type: Superiority; Unstratified HR = 0.32, 95% CI 2-sided [0.16 to 0.65] — Cox proportional hazard model. (HR < 1.0 indicates a lower average event rate and a longer survival for blinatumomab relative to HC3.)

4. Secondary Outcome: Percentage of Participants With an MRD Response Within 29 Days of Treatment Initiation
Description: At the end of the first treatment cycle (Day 29) a bone marrow aspiration/biopsy was performed and evaluated by the central MRD laboratory.
  MRD response was defined as MRD level < 10^-4, by polymerase chain reaction (PCR) or flow cytometry, at the end of treatment (Cycle 1 Day 29) with study drug. Participants who were part of the MRD Evaluable Set and were missing the end of treatment (Cycle 1 Day 29) assessment for a respective MRD assessment method were considered not to have achieved a response.
Time Frame: Up to End of Treatment (Cycle 1, Day 29)
Population: MRD Evaluable Set: participants for whom an evaluable baseline MRD marker can be found with either of the MRD assessment methods of PCR or flow cytometry.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HC3 Chemotherapy | Blinatumomab
Number analyzed (Participants) | 56 | 54
percentage of participants
  MRD Response by PCR: number analyzed (Participants) | 49 | 49
  MRD Response by PCR | 53.1 [38.3 to 67.5] | 93.9 [83.1 to 98.7]
  MRD Response by Flow Cytometry: number analyzed (Participants) | 55 | 54
  MRD Response by Flow Cytometry | 60.0 [45.9 to 73.0] | 92.6 [82.1 to 97.9]
Statistical Analysis 1: Comparison: HC3 Chemotherapy vs Blinatumomab; MRD response by PCR; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel test adjusting for the stratification factors: age (1 to 9 years vs other [< 1 year and > 9 years]), and marrow/MRD status (M1 with MRD level < 10^-3 vs M1 with MRD level ≥ 10^-3 vs M2)
Statistical Analysis 2: Comparison: HC3 Chemotherapy vs Blinatumomab; MRD response by flow cytometry; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel test adjusting for the stratification factors: age (1 to 9 years vs other [< 1 year and > 9 years]), and marrow/MRD status (M1 with MRD level < 10-3 vs M1 with MRD level ≥ 10-3 vs M2)

5. Secondary Outcome: Cumulative Incidence of Relapse (CIR)
Description: CIR estimate, presented as median months to relapse, calculated from date of achievement of first CR, using the cumulative incidence method (Fine JP, Gray RJ:1999). Deaths prior to relapse not considered related to an otherwise undocumented relapse were treated as a competing risk. Participants still alive without a date of relapse were censored at the time of last follow-up.
  Relapse=presence of ≥1 of the following:
  * isolated bone marrow relapse (M3 marrow [representative bone marrow aspirate or biopsy with ≥25% blasts] in the absence of extramedullary involvement)
  * combined bone marrow relapse (M2 [representative bone marrow aspirate or biopsy with ≥5% and <25% blasts] or M3 marrow and ≥1 extramedullary manifestation of acute lymphoblastic leukemia)
  * central nervous system extramedullary relapse
  * testicular extramedullary relapse
  * extramedullary relapse at other sites
  Months were calculated as days from randomization to event/censor date, divided by 30.5.
Time Frame: At final analysis, the overall maximum follow-up time was 82.0 months.
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | HC3 Chemotherapy | Blinatumomab
Number analyzed (Participants) | 57 | 54
months | 7.9 [5.8 to 18.6] | NA [NA to NA] — NA=not estimable (median CIR and confidence intervals were not reached at final analysis)
Statistical Analysis 1: Comparison: HC3 Chemotherapy vs Blinatumomab; Test type: Superiority; Hazard Ratio (HR) = 0.29, 95% CI 2-sided [0.16 to 0.52] — The subdistribution HR estimates are obtained from the subdistribution Cox model. (HR < 1.0 indicates a lower average event rate and a longer relapse-free time for blinatumomab relative to HC3.)
Statistical Analysis 2: Comparison: HC3 Chemotherapy vs Blinatumomab; Test type: Superiority; Stratified hazard ratio (HR) = 0.27, 95% CI 2-sided [0.15 to 0.48] — The subdistribution HR estimates are obtained from the subdistribution Cox model. (HR < 1.0 indicates a lower average event rate and a longer relapse-free time for blinatumomab relative to HC3.) Stratification factors are age and marrow/MRD status

6. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Related Adverse Events (TRAEs)
Description: Adverse event (AE): any untoward medical occurrence. Serious AE: an AE meeting at least 1 of the following serious criteria: fatal; life-threatening; requires in-patient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; congenital anomaly/birth defect; other medically important serious event. Severity was graded according to the Common Terminology Criteria for AEs (CTCAE) version 4.03: 1=mild, 2=moderate, 3=severe, 4=life-threatening, 5=death. Investigational product (IP) in the HC3 arm refers to dexamethasone, methotrexate, daunorubicin, erwinase, ifosfamide, asparaginase, and vincristine, and in the blinatumomab arm refers to blinatumomab. Treatment-related refers to the assessment of a relationship between IP and the event.
Time Frame: From first dose of IP through the last dose of IP (up to Day 29) plus 30 days.
Population: Safety Analysis Set: participants who received protocol-specified therapy analyzed according to the treatment they received.
Measure: Number; unit: participants
Arm/Group | HC3 Chemotherapy | Blinatumomab
Number analyzed (Participants) | 52 | 54
participants
  TEAEs | 50 | 54
  TEAEs Grade ≥ 3 | 43 | 33
  Serious TEAEs | 24 | 15
  Fatal TEAEs | 0 | 0
  TEAEs Leading to Discontinuation of IP | 0 | 2
  TEAEs Leading to Interruption of IP | 2 | 6
  TRAEs | 41 | 45
  TRAEs Grade ≥ 3 | 33 | 9
  Serious TRAEs | 15 | 9
  Fatal TRAEs | 0 | 0
  TRAEs Leading to Discontinuation of IP | 0 | 2
  TRAEs Leading to Interruption of IP | 2 | 5

7. Secondary Outcome: Number of Participants With TEAEs of Interest
Description: TEAEs of interest included capillary leak syndrome (CLS), cytokine release syndrome (CRS), decreased immunoglobulins (DI), elevated liver enzymes (ELE), embolic and thrombotic events (ETE), infections (INF), infusion reactions without considering duration (IRWCD), medication errors (ME), neurologic events (NE), neutropenia and febrile neutropenia (NFN), pancreatitis (PNC), tumor lysis syndrome, leukoencephalopathy, immunogenicity. Severity was graded according to the CTCAE version 4.03: 1=mild, 2=moderate, 3=severe, 4=life-threatening, 5=death.
Time Frame: From first dose of IP through the last dose of IP (up to Day 29) plus 30 days.
Population: Safety Analysis Set: who received protocol-specified therapy analyzed according to the treatment they received.
Measure: Number; unit: participants
Arm/Group | HC3 Chemotherapy | Blinatumomab
Number analyzed (Participants) | 52 | 54
participants
  CLS Events | 1 | 0
  CLS Events Grade ≥ 3 | 1 | 0
  Serious CLS Events | 1 | 0
  Fatal CLS Events | 0 | 0
  CLS Events Leading to Discontinuation of IP | 0 | 0
  CLS Events Leading to Interruption of IP | 0 | 0
  CRS Events | 1 | 2
  CRS Events Grade ≥ 3 | 0 | 0
  Serious CRS Events | 0 | 0
  Fatal CRS Events | 0 | 0
  CRS Events Leading to Discontinuation of IP | 0 | 0
  CRS Events Leading to Interruption of IP | 0 | 0
  DI Events | 6 | 9
  DI Events Grade ≥ 3 | 1 | 1
  Serious DI Events | 0 | 1
  Fatal DI Events | 0 | 0
  DI Events Leading to Discontinuation of IP | 0 | 0
  DI Events Leading to Interruption of IP | 0 | 0
  ELE Events | 15 | 7
  ELE Events Grade ≥ 3 | 9 | 3
  Serious ELE Events | 1 | 0
  Fatal ELE Events | 0 | 0
  ELE Events Leading to Discontinuation of IP | 0 | 0
  ELE Events Leading to Interruption of IP | 0 | 0
  ETE Events | 0 | 4
  ETE Events Grade ≥ 3 | 0 | 2
  Serious ETE Events | 0 | 0
  Fatal ETE Events | 0 | 0
  ETE Events Leading to Discontinuation of IP | 0 | 0
  ETE Events Leading to Interruption of IP | 0 | 0
  INF Events | 18 | 25
  INF Events Grade ≥ 3 | 6 | 11
  Serious INF Events | 6 | 4
  Fatal INF Events | 0 | 0
  IFN Events Leading to Discontinuation of IP | 0 | 0
  IFN Events Leading to Interruption of IP | 0 | 0
  IRWCD Events | 4 | 37
  IRWCD Events Grade ≥ 3 | 0 | 2
  Serious IRWCD Events | 0 | 1
  Fatal IRWCD Events | 0 | 0
  IRWCD Events Leading to Discontinuation of IP | 0 | 0
  IRWCD Events Leading to Interruption of IP | 0 | 0
  ME Events | 0 | 1
  ME Events Grade ≥ 3 | 0 | 0
  Serious ME Events | 0 | 1
  Fatal ME Events | 0 | 0
  ME Events Leading to Discontinuation of IP | 0 | 0
  ME Events Leading to Interruption of IP | 0 | 1
  NE Events | 15 | 26
  NE Events Grade ≥ 3 | 1 | 3
  Serious NE Events | 1 | 5
  Fatal NE Events | 0 | 0
  NE Events Leading to Discontinuation of IP | 0 | 2
  NE Events Leading to Interruption of IP | 1 | 3
  NFN Events | 28 | 12
  NFN Events Grade ≥ 3 | 27 | 11
  Serious NFN Events | 12 | 0
  Fatal NFN Events | 0 | 0
  NFN Events Leading to Discontinuation of IP | 0 | 0
  NFN Events Leading to Interruption of IP | 0 | 0
  PNC Events | 1 | 0
  PNC Events Grade ≥ 3 | 1 | 0
  Serious PNC Events | 1 | 0
  Fatal PNC Events | 0 | 0
  PNC Events Leading to Discontinuation of IP | 0 | 0
  PNC Events Leading to Interruption of IP | 0 | 0
  Tumour Lysis Syndrome Events | 0 | 0
  Leukoencephalopathy Events | 0 | 0
  Immunogenicity Events | 0 | 0

8. Secondary Outcome: Number of Participants With Shifts From Baseline Grade 0 or 1 to Worst Postbaseline Grade 3 or 4 Clinical Chemistry and Hematology Values
Description: Severity was graded according to the CTCAE version 4.03: 1=mild, 2=moderate, 3=severe, 4=life-threatening, 5=death. Increases (↑) or decreases (↓) in laboratory value grades (Gr) from baseline (BL) to worst postbaseline (→ PB) grade are presented. NA=not available.
Time Frame: Up to Day 29 (± 2 days).
Population: Safety Analysis Set: who received protocol-specified therapy analyzed according to the treatment they received.
Measure: Number; unit: participants
Arm/Group | HC3 Chemotherapy | Blinatumomab
Number analyzed (Participants) | 52 | 54
participants
  Potassium ↑ BL Gr 0 → PB Gr 3 | 0 | 1
  Potassium ↓ BL Gr 0 → PB Gr 3 | 4 | 5
  Potassium ↓ BL Gr 0 → PB Gr 4 | 1 | 1
  Albumin ↓ BL Gr 0 → PB Gr 3 | 0 | 1
  Calcium ↓ BL Gr 0 → PB Gr 4 | 1 | 1
  Alanine Aminotransferase ↑ BL Gr 0 → PB Gr 3 | 1 | 0
  Alanine Aminotransferase ↑ BL Gr 1 → PB Gr 3 | 9 | 5
  Aspartate Aminotransferase ↑ BL Gr NA → PB Gr 3 | 1 | 0
  Aspartate Aminotransferase ↑ BL Gr 0 → PB Gr 3 | 2 | 0
  Aspartate Aminotransferase ↑ BL Gr 1 → PB Gr 3 | 5 | 1
  Aspartate Aminotransferase ↑ BL Gr 1 → PB Gr 4 | 1 | 0
  Gamma-Glutamyl Transferase ↑ BL Gr NA → PB Gr 3 | 0 | 1
  Gamma-Glutamyl Transferase ↑ BL Gr 0 → PB Gr 3 | 3 | 4
  Gamma-Glutamyl Transferase ↑ BL Gr 1 → PB Gr 3 | 6 | 2
  Gamma-Glutamyl Transferase ↑ BL Gr 1 → PB Gr 4 | 0 | 3
  Amylase ↑ BL Gr 0 → PB Gr 3 | 1 | 1
  Amylase ↑ BL Gr 0 → PB Gr 4 | 1 | 0
  Amylase ↑ BL Gr 1 → PB Gr 3 | 0 | 1
  Lipase ↑ BL Gr 0 → PB Gr 3 | 3 | 2
  Lipase ↑ BL Gr 0 → PB Gr 4 | 1 | 2
  Bilirubin ↑ BL Gr 0 → PB Gr 3 | 2 | 1
  Bilirubin ↑ BL Gr 0 → PB Gr 4 | 1 | 0
  Creatinine ↑ BL Gr NA → PB Gr 3 | 0 | 2
  Hemoglobin ↓ BL Gr 0 → PB Gr 3 | 1 | 0
  Hemoglobin ↓ BL Gr 1 → PB Gr 3 | 4 | 1
  Platelets ↓ BL Gr 0 → PB Gr 3 | 7 | 6
  Platelets ↓ BL Gr 0 → PB Gr 4 | 13 | 6
  Platelets ↓ BL Gr 1 → PB Gr 3 | 1 | 2
  Platelets ↓ BL Gr 1 → PB Gr 4 | 8 | 2
  Leukocytes ↓ BL Gr 0 → PB Gr 3 | 2 | 0
  Leukocytes ↓ BL Gr 0 → PB Gr 4 | 4 | 0
  Leukocytes ↓ BL Gr 1 → PB Gr 3 | 4 | 4
  Leukocytes ↓ BL Gr 1 → PB Gr 4 | 7 | 1
  Neutrophils ↓ BL Gr 0 → PB Gr 3 | 4 | 11
  Neutrophils ↓ BL Gr 0 → PB Gr 4 | 23 | 3
  Lymphocytes ↑ BL Gr 0 → PB Gr 3 | 0 | 1
  Lymphocytes ↓ BL Gr 0 → PB Gr 3 | 1 | 3
  Lymphocytes ↓ BL Gr 0 → PB Gr 4 | 1 | 1
  Lymphocytes ↓ BL Gr 1 → PB Gr 3 | 0 | 1
  Lymphocytes ↓ BL Gr 1 → PB Gr 4 | 1 | 2

9. Secondary Outcome: Kaplan-Meier Estimate of 100-Day Mortality After Allogeneic Hematopoietic Stem Cell Transplantation (alloHSCT)
Description: The analysis of 100-day mortality after alloHSCT was assessed for participants who received an alloHSCT while in remission and did not receive any additional anti-leukemic treatment. 100-day mortality after alloHSCT was calculated relative to the date of alloHSCT.
  The 100-day mortality rate after alloHSCT was defined as the percentage of participants having died up to 100 days after alloHSCT, estimated using the estimated time to death in percent calculated by Kaplan-Meier methods. Participants still alive were censored at the date they were last known to be alive.
Time Frame: From the date of alloHSCT until death/censor date; median follow up time was 1742.0 days for blinatumomab and 1619.0 days for HC3.
Population: HSCT Analysis Set: participants who underwent an HSCT while in remission without any other anti-leukemic therapy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HC3 Chemotherapy | Blinatumomab
Number analyzed (Participants) | 39 | 51
percentage of participants | 5.1 [1.3 to 19.0] | 3.9 [1.0 to 14.8]

10. Secondary Outcome: Number of Participants With Anti-Blinatumomab Antibodies Postbaseline (Blinatumomab Arm Only)
Description: Participants receiving blinatumomab had blood samples analyzed for binding antibodies. Samples testing positive for binding antibodies were also tested for neutralizing antibodies.
  Participants who were binding antibody-positive or neutralizing antibody-positive post-baseline with a negative or no result at baseline are presented.
Time Frame: Day 1 to Day 29.
Population: Safety Analysis Set: participants who received protocol-specified therapy analyzed according to the treatment they received. Participants in the blinatumumab arm with a post-baseline result.
Measure: Number; unit: participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 52
participants
  Binding Antibody Positive | 0
  Neutralizing Antibody Positive | 0

11. Secondary Outcome: Pharmacokinetics: Concentration at Steady State (Css) (Blinatumomab Arm Only)
Time Frame: Day 1: at least 10 hours after infusion start and up to 24 hours; Day 15
Population: Pharmacokinetic (PK) Analysis Set: participants who received any infusion of blinatumomab and had at least one PK sample collected.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Blinatumomab
Number analyzed (Participants) | 45
pg/mL | 884 (969)

12. Secondary Outcome: Pharmacokinetics: Clearance (CL) (Blinatumomab Arm Only)
Time Frame: Day 1: at least 10 hours after infusion start and up to 24 hours; Day 15
Population: PK Analysis Set: participants who received any infusion of blinatumomab and had at least one PK sample collected.
Measure: Mean (Standard Deviation); unit: L/hr/m^2
Arm/Group | Blinatumomab
Number analyzed (Participants) | 45
L/hr/m^2 | 1.14 (0.836)

ADVERSE EVENTS:
Time Frame: All-cause mortality is reported from randomization through the end of study; the median overall follow-up time was 55.2 months. Treatment-emergent adverse events are reported from the first dose of IP through the last dose of IP (up to Day 29) plus 30 days.
Description: All-cause mortality is reported for all participants enrolled/randomized in the study. Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Arm/Group | HC3 Chemotherapy | Blinatumomab
All-Cause Mortality (participants affected / at risk) | 28/57 | 11/54
Serious Adverse Events (participants affected / at risk) | 24/52 | 15/54
Other Adverse Events (participants affected / at risk) | 48/52 | 54/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HC3 Chemotherapy (N=52) | Blinatumomab (N=54)
Febrile neutropenia (Blood and lymphatic system disorders) | 9 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 1
Pyrexia (General disorders) | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Herpes virus infection (Infections and infestations) | 0 | 1
Klebsiella infection (Infections and infestations) | 0 | 1
Perineal cellulitis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 | 0
Blood immunoglobulin G decreased (Investigations) | 0 | 1
Body temperature increased (Investigations) | 0 | 1
Lipase increased (Investigations) | 1 | 0
Neurological examination abnormal (Investigations) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 1
Neurological symptom (Nervous system disorders) | 0 | 2
Seizure (Nervous system disorders) | 0 | 2
Catheter placement (Surgical and medical procedures) | 0 | 1
Capillary leak syndrome (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Complication associated with device (General disorders) | 0 | 1
Engraftment syndrome (Immune system disorders) | 0 | 1
Laryngotracheitis obstructive (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Vulvitis (Infections and infestations) | 1 | 0
B precursor type acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HC3 Chemotherapy (N=52) | Blinatumomab (N=54)
Anaemia (Blood and lymphatic system disorders) | 24 | 13
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 3
Leukopenia (Blood and lymphatic system disorders) | 3 | 0
Neutropenia (Blood and lymphatic system disorders) | 13 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 11 | 4
Aplasia (Congenital, familial and genetic disorders) | 4 | 2
Abdominal pain (Gastrointestinal disorders) | 11 | 7
Abdominal pain upper (Gastrointestinal disorders) | 4 | 4
Constipation (Gastrointestinal disorders) | 7 | 5
Diarrhoea (Gastrointestinal disorders) | 9 | 12
Nausea (Gastrointestinal disorders) | 9 | 23
Oral pain (Gastrointestinal disorders) | 3 | 1
Stomatitis (Gastrointestinal disorders) | 27 | 11
Vomiting (Gastrointestinal disorders) | 11 | 17
Fatigue (General disorders) | 2 | 3
Mucosal inflammation (General disorders) | 4 | 9
Pyrexia (General disorders) | 10 | 43
Hypertransaminasaemia (Hepatobiliary disorders) | 4 | 1
Hypogammaglobulinaemia (Immune system disorders) | 2 | 6
Immunodeficiency (Immune system disorders) | 0 | 4
Nasopharyngitis (Infections and infestations) | 1 | 3
Paronychia (Infections and infestations) | 0 | 3
Rhinitis (Infections and infestations) | 5 | 1
Alanine aminotransferase increased (Investigations) | 7 | 4
Antithrombin III decreased (Investigations) | 3 | 1
Aspartate aminotransferase increased (Investigations) | 5 | 2
Fluid balance positive (Investigations) | 3 | 2
Neutrophil count decreased (Investigations) | 2 | 5
Platelet count decreased (Investigations) | 8 | 7
White blood cell count decreased (Investigations) | 1 | 4
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 2
Headache (Nervous system disorders) | 8 | 20
Tremor (Nervous system disorders) | 0 | 5
Agitation (Psychiatric disorders) | 1 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Erythema (Skin and subcutaneous tissue disorders) | 2 | 6
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 6
Rash (Skin and subcutaneous tissue disorders) | 5 | 7
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 3
Haematoma (Vascular disorders) | 3 | 1
Hypertension (Vascular disorders) | 4 | 7
Hypotension (Vascular disorders) | 4 | 6
Anal inflammation (Gastrointestinal disorders) | 2 | 4
Pain (General disorders) | 3 | 1
Hepatotoxicity (Hepatobiliary disorders) | 3 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2022-08-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT02393859/Prot_002.pdf
  • Statistical Analysis Plan (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/59/NCT02393859/SAP_001.pdf